CLINICAL TRIAL: NCT04737421
Title: A Prospective, Non-interventional, Clinical Study to Evaluate the Safety, Performance and Clinical Benefits of Implants With TiUltra Technology and Associated Prosthetic Components
Brief Title: A Clinical Study on Implants With TiUltra Technology and Associated Prosthetic Components
Status: Active, not recruiting | Type: Observational
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Other Study IDs: T-192
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Marginal Bone Level Change
Keywords: bone remodelling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1 (G1): NobelActive TiUltra implants (3.0, NP, RP, WP): Subjects will be enrolled into Group 1 and treated with NobelActive TiUltra implants, only if it is driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic.
  Interventions: Device: NobelActive TiUltra implant
- Group 2 (G2): NobelParallel CC TiUltra implants (NP, RP; WP): Subjects will be enrolled into Group 1 and treated with NobelParallel CC TiUltra implants, only if it is driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic.
  Interventions: Device: NobelParallel CC TiUltra implants
- Group 3 (G3): NobelReplace CC TiUltra implants (NP, RP): Subjects will be enrolled into Group 1 and treated with NobelReplace CC TiUltra implants, only if it is driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic.
  Interventions: Device: NobelReplace CC TiUltra implants
- Group 4 (G4): Nobel Biocare N1 TiUltra TCC implants (NP, RP): Subjects will be enrolled into Group 1 and treated with Nobel Biocare N1 TiUltra TCC implants , only if it is driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic.
  Interventions: Device: Nobel Biocare N1 TiUltra TCC implants

INTERVENTIONS:
Device: NobelActive TiUltra implant — Subjects will be enrolled and treated with one of the above groups as per the their clinical requirement and standard of care of the clinic.
  Groups: Group 1 (G1): NobelActive TiUltra implants (3.0, NP, RP, WP)
Device: NobelParallel CC TiUltra implants — Subjects will be enrolled and treated with one of the above groups as per the their clinical requirement and standard of care of the clinic.
  Groups: Group 2 (G2): NobelParallel CC TiUltra implants (NP, RP; WP)
Device: NobelReplace CC TiUltra implants — Subjects will be enrolled and treated with one of the above groups as per the their clinical requirement and standard of care of the clinic.
  Groups: Group 3 (G3): NobelReplace CC TiUltra implants (NP, RP)
Device: Nobel Biocare N1 TiUltra TCC implants — Subjects will be enrolled and treated with one of the above groups as per the their clinical requirement and standard of care of the clinic.
  Groups: Group 4 (G4): Nobel Biocare N1 TiUltra TCC implants (NP, RP)

SUMMARY:
This is a multicenter, prospective, non-interventional study in which a total of 1000 subjects in need of a single, multiple or full arch restoration in any region of the mouth (healed or extracted) will be treated in up to 30 study centers. The primary aim of this study is to demonstrate non-inferiority of all NobelBiocare TiUltra implants to historic data from NobelActive TiUnite coated implant in terms of marginal bone level change over 5 years after final prosthetic delivery. Eligible subjects who provide their informed consent for participation will be enrolled into one of four groups, each sized to 250 individuals. They will be treated with the corresponding implant system assigned to the group. The allocation into a certain group is only driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic. Each subject will be followed for 5 years after definitive prosthetic placement

DETAILED DESCRIPTION:
Primary Objective: The primary endpoint is to evaluate the change in the marginal bone level from definitive prosthetic placement (baseline) to the 5-year follow-up visit.

Secondary Objective:The secondary objectives of this clinical investigation are:

* To evaluate the change in the marginal bone level from definitive prosthetic placement (baseline) to 1-year and 3-years follow-up visits
* To demonstrate cumulative implant survival and success rates from definitive prosthetic placement to 5 years follow-up visit
* To demonstrate cumulative prosthetic survival and success rates to 5 years follow-up visit
* To evaluate soft tissue outcome (as measured by bleeding index, plaque index and gingival index) to 5 years from definitive prosthetic placement.
* To evaluate SADE, USADE, ADE and DD from implant insertion until 5 years follow-up visit.

Study design: This is a multicenter, prospective, non-interventional study in which a total of 1000 subjects in need of a single, multiple or full arch restoration in any region of the mouth (healed or extracted) will be treated in up to 30 study centers. The study devices are divided into four groups:

* Group 1 (G1): NobelActive TiUltra implants (3.0, NP, RP, WP)
* Group 2 (G2): NobelParallel CC TiUltra implants (NP, RP; WP)
* Group 3 (G3): NobelReplace CC TiUltra implants (NP, RP)
* Group 4 (G4): Nobel Biocare N1 TiUltra TCC implants (NP, RP)

Subjects will be consecutively included provided they meet all of the inclusion criteria and none of the exclusion criteria. Eligible subjects who provide their informed consent for participation will be enrolled into one of four groups, each sized to 250 individuals. They will be treated with the corresponding implant system assigned to the group. The allocation into a certain group is only driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic. Each subject will be followed for 5 years after definitive prosthetic placement . Possible dropouts and withdrawals, as well as possible serious adverse (device) events, will be carefully monitored during the entire study period

Sequence of treatment: As part of the screening process each subject will undergo a pre-treatment standard of care examination to record demographic characteristics and medical history. The subjects will be informed of the treatment possibilities according to clinic standard of care and about the study. Depending on the clinical indication, clinician preferences and desired esthetic solution the subject will be enrolled into one of the four previously described groups (G1 to G4). Implant surgery-, bone and tissue regenerative- and prosthodontic procedures shall be performed according to IFU and standard of care. Implants may be placed in either healed or extraction sites utilizing one-stage or two-stage surgical protocol with immediate, early or delayed loading to restore single missing tooth, partial or fully edentulous jaws. The treating clinician should decide individually when definitive prosthesis installation is suitable for each subject. Standard of care follow-up visits should be scheduled as close as possible to 1-, 3- and 5- years after definitive prosthetic placement, to ascertain a homogenous data set. Deidentified periapical radiographs from each subject visit shall be uploaded to the study eCRF. All images will be forwarded to the core lab for independent analysis. As part of the screening process each subject will undergo a pre-treatment standard of care examination to record demographic characteristics and medical history. The subjects will be informed of the treatment possibilities according to clinic standard of care and about the study.

Depending on the clinical indication, clinician preferences and desired esthetic solution the subject will be enrolled into one of the four previously described groups (G1 to G4). Implant surgery-, bone and tissue regenerative- and prosthodontic procedures shall be performed according to IFU and standard of care. Implants may be placed in either healed or extraction sites utilizing one-stage or two-stage surgical protocol with immediate, early or delayed loading to restore single missing tooth, partial or fully edentulous jaws. The treating clinician should decide individually when definitive prosthesis installation is suitable for each subject.

Study duration: Once the subject has provided written informed consent and fulfilled all inclusion and none of the exclusion criteria, he/she is considered enrolled. Subject enrolment period is expected to take 7 months from time of initiation at each site. Enrolment in each group will stop once the total group size of 250 subjects has been met. The clinical investigation will continue until each subject has been followed for 5-years after final prosthetic delivery.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed the informed consent
* Subject is between 18 and 70 years of age
* Subjects presented with the need of single, multiple or full arch implant rehabilitation in any region of the mouth.
* Subject with medical and anatomical conditions that are in accordance with the applicable instructions for use (IFU).
* Subject with sufficient bone volume for implant placement.
* Subject is compliant with good oral hygiene as judged by the clinician.

Exclusion Criteria:

* Anatomical conditions discovered during surgery preventing the use of intended implant system.
* Subjects with history of allergy or adverse reactions to any materials used
* Uncontrolled diabetes (subjects with history of diabetes mismanagement and/or known A1c level above 8%)*
* Heavy smokers (>10 cigarettes per day)
* Severe bruxism or dysfunctional tendencies
* Previous oro-maxillo facial radiotheraphy
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc)
* Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous radiation.
* Acute, untreated periodontitis in the planned implantation site or adjacent tissue.
* Infections in the planned implantation site or adjacent tissue.
* Documented complete remission of >3 years if history of non-oral cancer.
* Pregnant or lactating women at the time of implant insertion. *Assessment of A1C level is not required unless it is standard of care at the treating clinic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be consecutively included provided they meet all of the inclusion criteria and none of the exclusion criteria.They will be treated with the corresponding implant system assigned to the group. The allocation into a certain group is only driven by the subject's clinical and restorative requirement and standard of care at the enrolling study clinic. Each subject will be followed for 5 years after definitive prosthetic placement.
  If the subject wishes to withdraw from the clinical study, he/she may do so at any time and for any reason during the clinical study. If provided, the reason for withdrawal should be recorded and documented in the subject's medical record and in the eCRF.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level change | Definitive prosthetic delivery to 5-years follow-up
  The primary endpoint is to evaluate the change in the marginal bone level from definitive prosthetic placement (baseline) to the 5-year follow-up visit.

SECONDARY OUTCOMES:
Marginal bone level change | Definitive Prosthetic delivery to 1-year, Definitive Prosthetic delivery to 3-years
  To evaluate the change in the marginal bone level from definitive prosthetic placement (baseline) to 1-year and 3-years follow-up visits
Cumulative Survival rate/Cumulative success rate | Definitive prosthetic delivery to 5-year follow-up
  To demonstrate cumulative implant survival and success rates from definitive prosthetic placement to 5 years follow-up visit
Prsothetic suviival and success rate | Definitive prosthetic delivery to 5-years follow-up
  To demonstrate cumulative prosthetic survival and success rates to 5 years follow-up visit
Sost tissue outcome- Bleeding index | Definitive prosthetic delivery to 5-years follow-up
  To evaluate soft tissue outcome as measured by bleeding index from definitive prosthetic placement to 5 years follow-up visit
Sost tissue outcome- Plaque index | Definitive prosthetic delivery to 5-years follow-up
  To evaluate soft tissue outcome as measured by plaque index from definitive prosthetic placement to 5 years follow-up visit.
Sost tissue outcome- Ginigval index | Definitive prosthetic delivery to 5-years follow-up
  To evaluate soft tissue outcome as measured by gingival index from definitive prosthetic placement to 5 years follow-up visit
Adverse event | Implant insertion to 5-years follow-up
  To evaluate Serious Adverse Device Effects , Unanticipated Serious Adverse Device Effect , Adverse Device Effects and Device Deficiency from implant insertion until 5 years follow-up visit.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (5):
  - Madison Prosthodontics, Madison, Alabama
  - Northwest Oral and Maxillofacial Surgery, Arlington Heights, Illinois
  - Midwest Dental Implantology, Saint Charles, Illinois
  - New York Center for Orthognathic and Maxillofacial Surgery, New York, New York
  - Periodontal Associates, Tualatin, Oregon
- Australia (3):
  - Dentartisans Pty ltd, Pyrmont, New South Wales
  - Bc Prosthodontics, West Perth, Perth
  - Melbourne Dental School The University of Melbourne, Melbourne
- Austria (2):
  - Akademie für orale Implantologie GmbH & Co, Vienna
  - Implantologie und Ästhetische Zahnheilkunde, Vienna
- Herning Implantat Center, Herning, Herning, Denmark
- Dental Center Helmiäinen, Tampere, Finland
- France (3):
  - Cabinet du Dr Noharet, Lyon
  - BGLP, Montpellier
  - IFCIA, Paris
- DrS - Schöne Zähne - Dr. Scherg Praxis für Implantologie & Ästhetik, Karlstadt am Main, Germany
- Italy (2):
  - Studio Odontoiatrico Specialistico Ban Mancini Fabbri, Cattolica
  - UOC di Chirurgia Maxillo-Facciale e Odontoiatria, Verona
- Netherlands (3):
  - Staas & Bergmans Zorgvooruwmond B.V., 's-Hertogenbosch
  - ParoBrea- Parodontologie & Implantologie, Breda
  - Department of Oral and Maxillofacial Surgery University Medical Center Groningen, Groningen
- The Oris Dental Harstad, Harstad, Norway
- Maló Clinic, Lisbon, Portugal
- Spain (3):
  - Clinica Lluch, Barcelona
  - Clinica Dental Crooke & Laguna, Málaga
  - Altés & Mesquida, Palma de Mallorca
- Sweden (2):
  - Folktandvården Västra Götaland, Brånemarkkliniken, Gothenburg
  - Pequrio AB, Malmo
- Switzerland (4):
  - Dentalspecialist, Egerkingen
  - Brunner Praxis für Zahnmedizin, Lucerne
  - Centrella Zahnärzte, Oberrieden
  - Bodensee-Implantat-Zentrum AG, Rorschach

IPD SHARING:
Plan to Share IPD: No